CLINICAL TRIAL: NCT07215728
Title: Computational Analysis Using Machine Learning Algorithms of Electronic Medical Record Data From Patients With Osteosarcoma or Ewing's Sarcoma
Brief Title: Machine Learning Applied to EHRs Data of Patients With Sarcoma
Acronym: AMLAS
Status: Completed | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Collaborators: IRCCS Istituto Ortopedico Rizzoli di Bologna (Unknown)
Responsible Party: Sponsor
Other Study IDs: AMLAS2025; AMLAS2025 (Other: University of Milan-Bicocca)
Record Dates: First submitted 2025-10-02; First posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-09

CONDITIONS: Sarcoma; Osteosarcoma; Ewing Sarcoma
Keywords: sarcoma; osteosarcoma; Ewing sarcoma; machine learning; computational statistics
MeSH Terms: conditions — Sarcoma; Osteosarcoma; Sarcoma, Ewing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Osteosarcoma: Data of patients diagnosed with osteosarcoma
  Interventions: Other: No intervention studied
- Ewing sarcoma: Data of patients diagnosed with Ewing sarcoma
  Interventions: Other: No intervention studied

INTERVENTIONS:
Other: No intervention studied — No intervention studied

SUMMARY:
Application of computational statistics and machine learning methods to data derived from electronic health records of patients diagnosed with sarcoma.

DETAILED DESCRIPTION:
This observational, retrospective, multicenter study will be conducted on a group of patients treated at the Rizzoli Orthopedic Institute in Bologna and followed throughout their treatment. The study population includes patients of both sexes and all ages, affected by the two types of bone sarcoma typical of young people, with histologically confirmed diagnoses. The musculoskeletal tumors referred to in the study are osteosarcoma (OS) and Ewing's sarcoma (ES). Both are rare and very aggressive tumors, with a prognosis that remains unsatisfactory. These characteristics limit the possibility of conducting ad hoc studies on large case series that would allow the characterization of patients affected by these conditions in order to identify prognostic predictors. The clinical registries of specialized centers such as the Rizzoli Orthopedic Institute (IOR), which has always been a reference point for the diagnosis and treatment of sarcomas, are a source of very relevant data in this regard, allowing the collection of observational data gathered prospectively over time. The aim of this retrospective observational study is to characterize clusters of patients with different prognostic profiles and, secondarily, to identify the most predictive characteristics with respect to the prognosis of patients, applying computational intelligence algorithms using the open-source programming language R to already available data.

At the Simple Departmental Structure (SSD) of Anatomy and Pathological Histology of the Rizzoli Orthopaedic Institute (IOR), two datasets containing these variables are available and ready for use:

* patients diagnosed with osteosarcoma at the IOR between January 1, 2003, and December 31, 2012.
* patients diagnosed with Ewing's sarcoma at the IOR from 01/01/2003 to 31/12/2012.

Following ethical approval, access to these data will be requested, to be subsequently analyzed with computational intelligence algorithms (e.g., Random Forests) to determine the characteristics most predictive of prognosis (using a technique called "recursive feature elimination").

ELIGIBILITY:
Inclusion criteria: confirmed diagnosis of osteosarcoma or Ewing sarcoma between 2003 and 2012 at the IRCCS Rizzoli Orthopaedic Institute.

Exclusion criteria: diagnosis other than osteosarcoma or Ewing sarcoma and/or diagnosis made before 2003 and after 2012.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Information unavailable.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2003-01-01 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2012-12-31 (Actual)

PRIMARY OUTCOMES:
Survival | 6 months
  Survival of patients during the follow-up

IPD SHARING:
Plan to Share IPD: Undecided
If we have the authorization from the Ethical Committee of the IOR hospital, we might consider sharing the data in the future.

REFERENCES:
- [Background] Fernandes K, Chicco D, Cardoso JS, Fernandes J. Supervised deep learning embeddings for the prediction of cervical cancer diagnosis. PeerJ Comput Sci. 2018 May 14;4:e154. doi: 10.7717/peerj-cs.154. eCollection 2018. PMID 33816808
- [Background] Chicco D, Oneto L. Computational intelligence identifies alkaline phosphatase (ALP), alpha-fetoprotein (AFP), and hemoglobin levels as most predictive survival factors for hepatocellular carcinoma. Health Informatics J. 2021 Jan-Mar;27(1):1460458220984205. doi: 10.1177/1460458220984205. PMID 33504243
- [Background] Chicco D, Haupt R, Garaventa A, Uva P, Luksch R, Cangelosi D. Computational intelligence analysis of high-risk neuroblastoma patient health records reveals time to maximum response as one of the most relevant factors for outcome prediction. Eur J Cancer. 2023 Nov;193:113291. doi: 10.1016/j.ejca.2023.113291. Epub 2023 Aug 19. PMID 37708628
- [Background] Cerono G, Melaiu O, Chicco D. Clinical Feature Ranking Based on Ensemble Machine Learning Reveals Top Survival Factors for Glioblastoma Multiforme. J Healthc Inform Res. 2023 Sep 20;8(1):1-18. doi: 10.1007/s41666-023-00138-1. eCollection 2024 Mar. PMID 38273986
- [Background] Chicco D, Oneto L, Cangelosi D. DBSCAN and DBCV application to open medical records heterogeneous data for identifying clinically significant clusters of patients with neuroblastoma. BioData Min. 2025 Jun 12;18(1):40. doi: 10.1186/s13040-025-00455-8. PMID 40506780